CLINICAL TRIAL: NCT01880944
Title: Evaluation of Usefulness of Contrast Enhanced MRI in Evaluation of Spine Trauma: Prospective Study
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Guen Young Lee, Cinical assistant professor, Seoul National University Bundang Hospital
Other Study IDs: B-1304-199-003
Record Dates: First submitted 2013-06-14; First posted 2013-06-19 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Trauma
Keywords: spine; trauma; MRI; contrast
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ER-spine trauma: patients with spinal trauma, who initially visits in emergency room
  Interventions: Other: NC-MRI, CE-MRI
- OUT-spine trauma: patients with spinal trauma, who initially visits in outpatient clinic
  Interventions: Other: NC-MRI, CE-MRI

INTERVENTIONS:
Other: NC-MRI, CE-MRI — non-contrast spine MRI(NC-MRI) contrast-enhanced spine MRI(CE-MRI)
  Other Names: non-contrast spine MRI(NC-MRI); contrast-enhanced spine MRI(CE-MRI)

SUMMARY:
Non-contrast MRI with T2 fat suppression has been a useful imaging modality in evaluation spinal trauma.

However, the role of contrast enhancement has not investigated in patients with spinal trauma.

Therefore, this prospective study aims to evaluate the usefulness of contrast enhanced MRI for spinal trauma W/U clinically.

The study hypothesis is that there is no additional gain in addition of contrast enhanced study to routine non-contrast MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who provided the informed consent
2. Patients with spinal trauma
3. Patients with age of 19 years or more

Exclusion Criteria:

1. Relative contraindication of MR contrast

   * previous history of any adverse event after injection of magnetic resonance contrast
   * pregnant or breast-feeding state
   * within 2 weeks after liver transplantation
   * epileptic disorder
2. Patients impossible with follow-up period of at least 2 months clinically
3. Patients with severely impaired renal function of estimated glomerular filtration rate (GFR) < 30 mL/min/1.73m2 and/or on dialysis
4. patients with age less than 19 years

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 patients that fulfilled the following criteria
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-06-24 (Actual); Primary Completion 2016-12-14 (Actual); Study Completion 2017-02-14 (Actual)

PRIMARY OUTCOMES:
The rate (%) of change of treatment option between non-surgery vs. surgery, after review of enhanced MRI finding, compared with non-enhanced MRI only | 2 months
  The rate (%) of change of treatment option between non-surgery vs. surgery, after review of enhanced MRI finding, compared with non-enhanced MRI only
Confidence level | 2 months
  Confidence level (1, definitely negative; 2, probably negative; 3, equivocal; 4, probably positive; 5, definitely positive) for lesion of spinal body, posterior compartment, soft tissue (posterior ligamentous complex of thoracolumbar spine and discoligamentous complex of cervical spine), spinal cord, and epidural/subdural hematoma/hemorrhage

SECONDARY OUTCOMES:
Diagnostic accuracy of non-enhanced and enhanced MRI | 2 months
  Diagnostic accuracy of non-enhanced and enhanced MRI in patients with operations for each anatomical lesion (e.g. fracture of body, fracture of posterior compartment, soft tissue injury, cord injury, and epidural/subdural hematoma)
Inter- and intra-reader agreement of confidence level | 2 months
  Inter- and intra-reader agreement of confidence level between non-enhanced and enhanced MRI

OTHER OUTCOMES:
Prognostic value of enhanced MRI | 2 months
  Prognostic value of enhanced MRI, compared with non-enhanced MRI, based on clinical feature during follow-up period: TLICS(thoracolumbar injury classification and severity score) or SLIC(subaxial cervical injury classification system)score for non-surgery group vs. surgery group
The rate (%) of change of treatment plan | 2 months
  The rate (%) of change of treatment plan between posterior vs. anterior vs. anterior & posterior approaches, after review of enhanced MRI finding, compared with non-enhanced MRI only

CONTACTS AND LOCATIONS:
Overall Officials: Guen Young Lee, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (2):
- South Korea (2):
  - Guen Young Lee, Seongnam-si, Gyenggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do